CLINICAL TRIAL: NCT05714592
Title: Evaluation of Optical Genome Mapping in Phi Negative Myeloproliferative Neoplasia in the Detection of Acquired Cytogenetic Abnormalities
Acronym: MYELOCARTOCH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Hôpital Jeanne de Flandre LIlle (Unknown); Centre Henri Becquerel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PI2022_843_0023
Record Dates: First submitted 2023-01-27; First posted 2023-02-06 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Myeloproliferative Neoplasm; Optical Genome Mapping; Cytogenetics; Clonality; Prognostic Stratification
Keywords: Myeloproliferative Neoplasm; Optical genome mapping; Cytogenetics; Clonality; Prognostic stratification
MeSH Terms: conditions — Myeloproliferative Disorders | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Optical genome mapping (Experimental)
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — The referring haematologist will suggest that the patient participate in the study during the consultation. In these patients, the investigators will perform OGM on the cytogenetic sample

SUMMARY:
Standard cytogenetics (CBA +/- FISH) is of diagnostic and prognostic interest in Ph- MPN. However, its value is limited by the low frequency of detected abnormalities. The development of tools to increase the sensitivity of detection of chromosomal alterations is therefore particularly adapted to these pathologies. Optical genome mapping (OGM) is a high resolution "long read" technique that allows the identification of structural and copy number variations at the whole genome level. Several recent studies suggest that OGM is a future tool for cytogenetic characterization of haematological disorders. Its ability to describe structural abnormalities, including balanced ones, represents a major advantage over currently used technologies. Thus, OGM seems to be the key tool for cytogenetics of haematological malignancies in the coming years, making it possible to replace, under certain conditions, not only karyotype and FISH, but CMA and even RT-MLPA for the search for fusion transcripts, thus filling in the gaps in these techniques while maintaining their advantages.

To define the place of this technology in Ph- MPN, the investigators will perform a OGM analysis on patients with Ph-MPN for whom bone marrow exploration is scheduled. These results will be compared with those of standard cytogenetics (CBA +/- FISH).

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years of age or older
* Diagnosis or follow-up of polycythemia vera, essential thrombocythemia or primary or secondary myelofibrosis
* Requires bone marrow cytogenetics at diagnosis or follow-up
* Understanding of the French language
* Information of the patient and collection of no objection
* Person affiliated to a social security regime

Exclusion Criteria:

* Patient with BCR::ABL positive myeloproliferative neoplasia.
* Person with a medical history that may impair the ability to understand the information notice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-01-27 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with the same abnormalises detected with both OGM and standard cytogenetics | one year
  Number of patients for whom the OGM finds at least the abnormalises detected by standard cytogenetics.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire d'Amiens, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No